CLINICAL TRIAL: NCT04066985
Title: Targeting Adolescent Depressive Symptoms: Effects of Two Single-Session, Online Interventions
Brief Title: Targeting Adolescent Depressive Symptoms Via Brief, Web-Based Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Child Mind Institute (Other)
Collaborators: Stony Brook University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00034009
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Depression; Depressive Disorder; Behavioral Symptoms; Mood Disorders; Mental Disorders
Keywords: Depression; Adolescent; Therapeutics; Mental Health
MeSH Terms: conditions — Depression; Depressive Disorder; Behavioral Symptoms; Mood Disorders; Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: All adolescent participants will be provided a study identifier and prompted to complete self-report questionnaires. Subsequently, a random number generator (embedded within Mindlogger, a Child Mind Institute developed data collection application) will be used to assign participants to one of three intervention conditions.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Neither investigators, outcomes assessor, youth, nor parents will know the condition assigned to the youth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Growth Mindset Intervention (Experimental): Includes one online, single-session program, the Growth Mindset Program. The 30-minute, self-administered youth program includes: An introduction to the brain and a lesson on neuroplasticity; Testimonials from older youths who describe their views that traits are malleable, due to the brain's plasticity; Further stories by older youths, describing times when they used "growth mindsets" to persevere during social/emotional setbacks; Study summaries noting how/why personality can change; And an exercise in which youths write notes to younger students, using scientific information to explain people's capacity for change.
  Interventions: Behavioral: Growth Mindset Online Single-Session Program
- Self-Kindness Intervention (Experimental): Includes one online, single-session program, the Self-Kindness Program. The 30-minute, self-administered youth program includes: An introduction to the science behind why adolescents might think disliking themselves is necessary for success and thus fear self-compassion; Scientific evidence and testimonials from other teens that being self-compassionate actually predicts being more successful socially and academically; Evidence-based tips for overcoming common, fear of self-compassion based obstacles to self-compassion in day to day life; And an exercise in which youths write notes to younger students, using scientific information to explain the benefits of using self-kindness.
  Interventions: Behavioral: Self-Kindness Online Single-Session Program
- Supportive Therapy Intervention (Active Comparator): Includes one online, single-session active comparator program, the Supportive Therapy Intervention. The ST SSI is designed to control for nonspecific aspects of intervention, including engagement in a computer program. The 30-minute, self-administered control group program includes: vignettes written by older youths who describe times when they benefited from sharing their feelings with friends or family; the same number of reading and writing activities as the web-based growth mindset intervention. However, the only goals of the ST intervention are to encourage youths to identify and express feelings to close others; the intervention does not teach or emphasize specific skills or beliefs.
  Interventions: Behavioral: Supportive Therapy Online Single-Session Program (Control)

INTERVENTIONS:
Behavioral: Growth Mindset Online Single-Session Program — 30minute self-administered program for youths
  Other Names: Project Personality
  Arms: Growth Mindset Intervention
Behavioral: Self-Kindness Online Single-Session Program — 30minute self-administered program for youths
  Other Names: Teenage Goals Project
  Arms: Self-Kindness Intervention
Behavioral: Supportive Therapy Online Single-Session Program (Control) — 30minute self-administered active comparator program for youths
  Other Names: Share Your Feelings Program
  Arms: Supportive Therapy Intervention

SUMMARY:
Major depression (MD) in youth is a serious psychiatric illness with extensive morbidity and mortality. The American Academy of Pediatrics recently released practice guidelines promoting primary care (PC)-based youth MD screening; however, even when diagnosed by PC providers, <50% of youth with MD access treatment. Thus, a need exists for interventions that are feasible for youths and parents to access and complete-and that may strengthen parents' likelihood of pursuing longer-term services. Single-session interventions (SSIs) may help forward these goals. SSIs include elements of comprehensive treatments, but their brevity makes them easier to disseminate at scale. Meta-analytic evidence suggests SSIs can reduce youth psychopathology, including self-administered (e.g., online) SSIs. One computer-based SSI, teaching growth mindset (GM; viewing personal traits as malleable), has reduced adolescent depressive symptoms in multiple RCTs. A second computer-based SSI was recently developed to reduce youth depressive symptoms via targeting reductions in self-hate-a symptom identified as important for the maintenance of other depressive symptoms in teenagers. This study will test whether either the growth mindset SSI (GM-SSI), the self-kindness SSI (SK-SSI), or both SSIs reduce symptoms of depression in adolescents, relative to an active "supportive therapy" SSI, which teaches adolescents to share their emotions with trusted others. Youths participating in existing research through the Healthy Brain Network (N=501) will receive either the growth mindset SSI (GM-SSI), the self-kindness SSI (SK-SSI), or the supportive therapy SSI (ST-SSI). The investigators will examine whether the GM-SSI and/or the SK-SSI, versus the ST-SSI will reduce youth depressive symptoms across three months. Results may identify two novel, potent, and brief interventions for adolescent depressive symptoms.

DETAILED DESCRIPTION:
Major depression (MD) is the leading cause of disability in youth, with a global economic burden of >$210 billion annually (Whiteford et al., 2013). However, up to 70% of youth with MD do not receive services (Vitiello et al., 2011). Even among those who do access treatment, 30-65% fail to respond (March et al, 2007), demonstrating a significant need for more potent, accessible interventions for adolescent depressive symptoms and disorders.

The goal of this project is to assess the acceptability and effectiveness of two computerized, single-session interventions that may reduce depressive symptoms in adolescents. Single-session interventions (SSIs) have shown promise in preventing and reducing youth mental health problems (see Schleider & Weisz, 2017, for a meta-analysis). The present trial will be the first to evaluate the effectiveness of two distinct SSIs, targeting different types of depressive symptoms, in comparison to an active, previously-established comparison intervention.

The first SSI is designed to instill a growth mindset in youth: the belief that personal behaviors and characteristics, such as depressive symptoms, are malleable rather than fixed (Schleider, Abel, & Weisz, 2015). In previous trial, a single-session growth mindset intervention significantly reduced depressive symptoms in high symptom-adolescents (Schleider & Weisz, 2018); however, questions still remain about the benefits of this intervention across all adolescents.

The second SSI, which has not been tested previously, is designed to strengthen self-kindness and reduce self-hate. This SSI targets self-hate because it is a symptom of depression that has been identified as especially "central," or more important to the maintenance of other kinds of depressive symptoms, in adolescents at-risk for emotional difficulties. Because self-hate is an especially central symptom, an SSI that systematically, precisely reduces it may serve as an especially potent intervention.

This study will test whether either the growth mindset SSI (GM-SSI), the self-kindness SSI (SK-SSI), or both reduces symptoms of depression in adolescents, relative to an active "supportive therapy" SSI, which teaches adolescents to share their emotions with trusted others (Schleider & Weisz 2018). Our second goal is to evaluate whether the GM-SSI and SK-SSI target and specifically improve proximal targets, unique to each SSI, immediately after SSI administration, relative to the comparison intervention (e.g., whether the GM-SSI improves perceived control relative to the comparison intervention, and whether the SK-SSI alters fear of self-compassion relative to the comparison intervention). To test these possibilities, adolescents recruited from the Healthy Brain Network research study (Advarra Pro00012309) (N=501, 167 per SSI condition; ages 11-17) will be randomized to one of three intervention conditions: the web-based GM-SSI; the web-based SK-SSI; or the web-based, supportive therapy (control) SSI, which has been validated previously (Schleider & Weisz, 2016; Schleider & Weisz, 2018). Adolescents will report on their depression symptoms, perceived control, self-compassion, and related domains of functioning at pre-intervention, post-intervention, and at three-month follow-up. The investigators predict the growth mindset and self-kindness web-based interventions will both lead to larger reductions in adolescent depression symptoms relative to the control intervention. Additionally, the investigators predict that the growth mindset SSI will lead to larger reductions in perceived control than the supportive therapy intervention, and that the self-kindness SSI will lead to larger reductions in fear of self-compassion relative to the control program. Results may identify two novel, potent, and brief interventions for adolescent depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Brain Network study participants
* Between the ages of 11-17 (inclusive)
* Fluent in English

Exclusion Criteria:

* Youth with parent-reported intellectual disability

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 501 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Mood and Feelings Questionnaire; Youth-Report | [Baseline to 3-month follow-up.]
  Youth-report measure of youth depressive symptoms. Youth rate 33 items reflecting internalizing symptoms on a 0-2 scale. Scores range from 0-66, with higher scores indicating greater symptom severity.

SECONDARY OUTCOMES:
Change in Screen for Child Anxiety and Related Disorders; Youth-Report | Baseline to 3-month follow-up.
  Youth-report measure of youth anxiety symptoms. Youth rate 41 items reflecting anxiety symptoms on a 0-2 scale. Scores range from 0-82, with higher scores indicating greater symptom severity.
Change in Implicit Theories of Personality Questionnaire; Youth-Report | Baseline to post-intervention; baseline to 3-month follow-up.
  Youth rate their agreement with 3 statements linked to the malleability of personality (e.g. "Your personality is something about you that you can't change very much"), on a 1-6 scale. Higher mean scores on these three items indicate a stronger fixed personality mindset, a lower scores, a stronger growth personality mindset (range: 1-6).
Change in Self-Hate Scale; Youth-Report | Baseline to post-intervention; baseline to 3-month follow-up.
  Youth rate 7 items evaluating the degree of their self-dislike (e.g., "I am ashamed of myself") on a 1-7 scale, with higher scores indicating greater levels of self-hate (possible score range: 7-49).
Change in Self-Judgment Subscale of Self-Compassion Scale; Youth-Report | Baseline to post-intervention; baseline to 3-month follow-up.
  Youth rate their agreement with 5 items reflecting self-judgment (e.g., "When times are really difficult, I tend to be tough on myself") on a 1-5 scale. These 5 items are a subscale within the Self-Compassion Scale, a 26-item self-report questionnaire measuring the six components of self-compassion (of which self-judgment is one). A mean is computed across responses to all 5 items to form a total Self-Judgment score (range: 1 to 5).
Change in Fear of Self-Compassion Scale; Youth-Report | Baseline to post-intervention; baseline to 3-month follow-up.
  Youth rate 15 items reflecting their level of fear about acting or thinking compassionately toward the self (e.g., 'I worry that if I start to develop compassion for myself I will become dependent on it') on a 0-4 scale. Scores range from 0-60.
Change in Beck Hopelessness Scale-Short Version; Youth-Report | Baseline to post-intervention; baseline to 3-month follow-up.
  Youth rate their agreement on 4 items reflecting their degree of hopelessness (e.g. "My future seems dark to me"), on a 0-3 scale. This 4-item scale is a shortened version of the 20-item Beck Hopelessness Scale designed for brief psychological screening purposes. Scores on the 4-item short version range from 0-12, with higher scores indicating higher levels of youth hopelessness.
Change in Primary Perceived Control Scale for Children; Youth-Report | Baseline to post-intervention; baseline to 3-month follow-up.
  Youth rate their agreement with 24 items reflecting their perceived ability to influence or alter objective events or conditions through personal effort (e.g., "I can do well on tests if I study hard") on a 0-3 scale. Scores range from 0-72, with higher scores indicating greater primary perceived control.
Change in Secondary Perceived Control Scale for Children; Youth-Report | Baseline to post-intervention; baseline to 3-month follow-up.
  Youth rate agreement with 20 items reflecting perceived ability to shape the personal impact of objective conditions on oneself, by adjusting oneself to fit those conditions (e.g. "When something bad happens, I can find a way to think about it that makes me feel better") on a 0-3 scale. Scores range from 0-60, with higher scores indicating greater secondary perceived control.

OTHER OUTCOMES:
Program Feedback Scale | Immediately post-intervention (0 - 2 minutes following the intervention)
  Youth rate agreement with 7 items reflecting their experience with the intervention to which they were assigned (e.g. "I enjoyed the program") on a 1-5 scale. Youth will be asked to complete a series of open-ended questions regarding their opinions about the program (e.g. "What did you like about the program? Please share as many true thoughts and feelings as you would like!").

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay M Alexander, MPH, Study Director — Child Mind Institute
Locations (1):
- Child Mind Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual-level participant data will be made publicly available in two databases: (1) COllaborative Informatics and Neuroimaging Suite (COINS), a HIPAA-compliant, open-source information system; (2) Longitudinal Online Research and Imaging System (LORIS), a HIPAA-compliant, web-based data and project management software. IPD associated with this project will be released to project collaborators upon the completion of the study (October 31, 2020). IPD associated with this project will be released to outside researchers at the next Healthy Brain Network quarterly data-release after the study's completion on October 31, 2020.
Supporting Information: Study Protocol
Time Frame: Protocol is outlined in this ClinicalTrials pre-registration. Statistical analysis plan will be uploaded to Open Science Framework prior to the study's onset October 31, 2019.
Access Criteria: Study protocol information is publicly available on clinicaltrials.gov. Statistical analysis plan will be made publicly available on Open Science Framework. IPD will be made publicly available on COINS and LORIS, and access to these databases requires a data usage agreement signed by the institution using the data.

REFERENCES:
- [Background] Schleider JL, Weisz JR. Little Treatments, Promising Effects? Meta-Analysis of Single-Session Interventions for Youth Psychiatric Problems. J Am Acad Child Adolesc Psychiatry. 2017 Feb;56(2):107-115. doi: 10.1016/j.jaac.2016.11.007. Epub 2016 Nov 25. PMID 28117056
- [Background] Schleider JL, Abel MR, Weisz JR. Implicit theories and youth mental health problems: a random-effects meta-analysis. Clin Psychol Rev. 2015 Feb;35:1-9. doi: 10.1016/j.cpr.2014.11.001. Epub 2014 Nov 7. PMID 25462109
- [Background] Schleider J, Weisz J. A single-session growth mindset intervention for adolescent anxiety and depression: 9-month outcomes of a randomized trial. J Child Psychol Psychiatry. 2018 Feb;59(2):160-170. doi: 10.1111/jcpp.12811. Epub 2017 Sep 18. PMID 28921523
- [Background] Schleider JL, Weisz JR. Reducing risk for anxiety and depression in adolescents: Effects of a single-session intervention teaching that personality can change. Behav Res Ther. 2016 Dec;87:170-181. doi: 10.1016/j.brat.2016.09.011. Epub 2016 Sep 26. PMID 27697671